CLINICAL TRIAL: NCT05638334
Title: An Open Label, Multicentre, Positron Emission Tomography (PET) Imaging Study Using Zirconium-89 to Investigate the Biodistribution and Tumour Uptake of a PD-L1x4-1BB Bispecific Antibody (S095012) in Patients With Advanced Solid Tumours
Brief Title: Immuno-positron Emission Tomography Study of 89Zr-S095012 in Patients With Advanced Solid Tumours
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL1-95012-002; 2021-001764-20 (EudraCT Number)
Record Dates: First submitted 2022-10-28; First posted 2022-12-06 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 89Zr-S095012 tracer with S095012 (Experimental)
  Interventions: Drug: 89Zr-S095012 tracer and S095012 will be administered via an IV infusion

INTERVENTIONS:
Drug: 89Zr-S095012 tracer and S095012 will be administered via an IV infusion — Imaging period 1 (Part A and Part B): The tracer will be administered with S095012 at non-therapeutic mass dose. The optimal mass dose of S095012 will be investigated in part A, and used in part B.
  Treatment period (Part A to C): S095012 will be administered with multiple 28 days- cycles in a Q2W schedule.
  Imaging period 2 (Part C): A second tracer dose will be administered at 1st treatment dose of S095012 in part C.

SUMMARY:
The purpose of this study is to assess the whole-body biodistribution and tumour uptake of 89Zr-S095012 in participants with solid tumours treated with S095012 (PD-L1x4-1BB bispecific antibody)

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of unresectable, locally advanced or metastatic solid tumour, for which standard treatment options are not available, no longer effective, or not tolerated
* At least one measurable target lesion as per RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Royal Marsden Prognosis score of 0 to 1 (score based on lactate dehydrogenase (LDH) value, albumin value and number of sites of metastasis)
* Adequate organ function as assessed by laboratory tests (especially adequate hepatic function)
* Negative test results for cytomegalovirus (CMV), Epstein-Barr virus (EBV), Hepatitis B virus (HBV), and Hepatitis C virus (HCV) infection, according to local standards.

Exclusion Criteria:

* Participants with no available archived material and no tumour lesions amenable to biopsy
* Participants with primary central nervous system malignancies, with Child-Pugh Class B8 or higher, or C liver cirrhosis
* Participants with active auto-immune disease or immune-related adverse event currently requiring systemic anti-inflammatory agent (more than 10mg/day prednisone or equivalent)
* Participants with a history of an opportunistic infection within a year before the administration of first study drug dose are excluded.
* Participants who received either systemic corticosteroids (> 10 mg per day of prednisone or equivalent) or other immunosuppressive medication during the 2 months prior to the first dose of the study drug are excluded.
* Participants with prior history of Grade ≥ 3 immune-related pneumonitis, colitis, hepatitis, or myocarditis
* Participants with a history of progressive multifocal leukoencephalopathy
* Participants must not have a history of active tuberculosis requiring treatment within 3 years prior to the start of treatment or a suspicion of latent tuberculosis by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Change in PET/CT scan images | Within 14 days following the tracer injection and baseline (before the first treatment administration (during the dose range finding period))
  Visual analysis of target lesions
Change in PET/CT scan images | Within 14 days following the tracer injection and baseline (before the first treatment administration)
  Visual analysis of target lesions
PET/CT scan images | Up to 8 days following the first treatment administration
  Visual analysis of target lesions
Parameters derived from PET scans for organs and tumour lesions | Within 14 days following the tracer injection and baseline (before the first treatment administration (during the dose range finding period))
  Change in Volume of interest
Parameters derived from PET scans for organs and tumour lesions | Within 14 days following the tracer injection and baseline (before the first treatment administration)
  Change in Volume of interest
Parameters derived from PET scans for organs and tumour lesions | Up to 8 days following first treatment administration
  Volume of interest
Parameters derived from PET scan images to assess uptake in tumour lesions and normal tissues | Within 14 days following the tracer injection and baseline (before the first treatment administration (during the dose range finding period))
  Change in Standardised uptake value (SUV)
Parameters derived from PET scan images to assess uptake in tumour lesions and normal tissues | Within 14 days following the tracer injection and baseline ( before the first treatment administration)
  Change in Standardised uptake value (SUV)
Parameters derived from PET scan images to assess uptake in tumour lesions and normal tissues | Up to 8 days following first treatment administration
  Standardised uptake value (SUV)
Serum PK parameters of 89Zr-S095012 during the range finding period (Part A) | radioactive plasma samples taken at : 5, 30, 60, 120 minutes, 6 hours (on Day-14) and on Day-13, Day-12, Day-10 and Day-7 following the tracer injection and before the first treatment administration (during the dose ranging period)
  Area under the curve (AUC)
Serum PK parameters of 89Zr-S095012 at baseline (Part B) | radioactive plasma samples taken at : 5, 30, 60, 120 minutes, 6 hours (on Day-14) and on Day-13, Day-12, Day-10 and Day-7 following the tracer injection and before the first treatment administration
  Area under the curve (AUC)
Serum PK parameters of 89Zr-S095012 on treatment (Part C- schedule 1) | radioactive plasma samples taken at : 5, 30, 60, 120 minutes, 6 hours (on Day 1) and on Day 2, Day 3, Day 5 and Day 8 following the first treatment administration
  Area under the curve (AUC)
Change in Comparison of 89Zr-S095012 tumour uptake (as described using Standardised Uptake Value and concentrations) before and on treatment with different doses of S095012. | In Part C (imaging period 2) between Day 1 and Day 8 of cycle 1 (the duration of cycle 1 is 28 days)
Incidence and severity of adverse events | Throughout the study up to 30 days after the last IMP for all AEs, or up to 90 days for all AEs related to the IMP and death
Number of patients discontinuing study intervention due to an adverse event | Throughout the study up to 30 days after the last IMP for all AEs, or up to 90 days for all AEs related to the IMP and death

SECONDARY OUTCOMES:
Serum PK parameters of S095012 during the range finding period (Part A) | plasma samples taken at : 5, 30, 60, 120 minutes, 6 hours (on Day-14) and on Day-13, Day-12, Day-10 and Day-7 following the tracer injection and before the first treatment administration (during the dose ranging period)
  Area under the curve (AUC)
Serum PK parameters of S095012 at baseline (Part B) | plasma samples taken at : 5, 30, 60, 120 minutes, 6 hours (on Day-14) and on Day-13, Day-12, Day-10 and Day-7 following the tracer injection and before the first treatment administration
  Area under the curve (AUC)
Serum PK parameters of S095012 on treatment (Part C - schedule 1) | plasma samples taken at : 5, 30, 60, 120 minutes, 6 hours (on Day 1) and on Day 2, Day 3, Day 5, Day 8 and Day 15 following the first treatment administration
  Area under the curve (AUC)
Organ and whole-body radiation exposure (milliSilvert per Mega Becquerel (mSv/MBq): Effective dose per organ and whole-body effective dose. | In Part A, B and C (imaging period 1) at Day-14
Preliminary antitumour activity assessment of S95012 | The events to be studied are Complete Response or Partial Response, from the first treatment administration up to one year (for patients with confirmed Complete response) or 2 years (for Patients with confirmed Partial Response).
  Percentage of patients who achieved complete response or partial response (ie, objective response rate (ORR)) according to Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1 (V1.1)

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Gronningen Oncologie, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier.
  * with a first patient enrolled as of 1 January 2004 onwards.
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com/

REFERENCES:
- See also: Find Results on Servier Clinical Trial Data website — http://clinicaltrials.servier.com/